CLINICAL TRIAL: NCT06795828
Title: The Effect of Emotional Support Given During Cesarean Section on Pain, Anxiety, and Surgical Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Assoc. Prof. Dr., Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TR SİVAS 06
Record Dates: First submitted 2025-01-13; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2023-07

CONDITIONS: Emotional Support During Cesarean Delivery
Keywords: Caesarean; Emotional Support; Pain; Anxiety; Fear of Surgery
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Providing emotional support during a caesarean section (Experimental): Empathetic approach, listening to the feelings and thoughts, welcoming the woman's behavior and expressions, telling her that she is breathing correctly, etc.), not judging the woman, being honest, using a soft and calm tone of voice, taking the baby or asking her opinion, encouraging her to endure the birth process, touching the woman and making physical contact, allowing her to practice her beliefs, showing the baby to the mother as soon as it is born and placing it in her arms.
  Interventions: Behavioral: Emotional support group
- Standard of care Group (No Intervention): The control group did not receive any treatment. Only Visual Analog Scale, State Anxiety Inventory and Surgical Fear Scale were applied (pre-test, post-test)

INTERVENTIONS:
Behavioral: Emotional support group — Women who met the inclusion criteria and volunteered to participate in the study and were provided emotional support were administered the Personal Information Form, Visual Analog Scale, State Anxiety Inventory and Surgical Fear Scale via face-to-face interview method on the first day of their hospitalization before the caesarean section (pre-test). This application lasted 15-20 minutes. Enter a brief, descriptive title for this arm of the study.
  Arms: Providing emotional support during a caesarean section

SUMMARY:
The study was conducted to determine the effect of emotional support given during cesarean section on pain, anxiety and surgical fear.

DETAILED DESCRIPTION:
The experimental study sample consisted of 120 women (emotional support group: 60, control group: 60). Data were collected using the Personal Information Form, Visual Analog Scale, State Anxiety Inventory and Surgical Fear Scale. In the comparison between the groups in the study, it was found that there was a statistically significant difference between the mean Visual Analog Scale scores of the women in the experimental and control groups in the pre-test (p<0.05), and no difference in the post-test (p˃0.05). In the post-test measured after emotional support, it was found that there was a statistically significant difference between the State Anxiety Inventory scores, short-term, long-term and total Surgical Fear Scale scores between the groups (p˂0.05). After emotional support, women's pain levels increased, anxiety and surgical fear levels decreased and their satisfaction with emotional support during birth increased. Women who did not receive emotional support had significantly increased pain, anxiety and surgical fear levels.

ELIGIBILITY:
Inclusion Criteria:

* Women who had a history of spinal anesthesia for the first time during a cesarean delivery,
* Who were going to have a planned cesarean before spontaneous contractions started,
* Who had no health problems with their babies,
* Who had no physical or mental problems themselves,
* Who had no communication difficulties,
* Women who volunteered to participate were included in the study.

Exclusion Criteria:

* Women who had a normal spontaneous delivery,
* Women who had a cesarean after labor/spontaneous contractions started,
* Women who had any health problems with their babies,
* Women who had a physical or mental illness themselves,
* Women who did not want to participate in the study were not included in the study.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Surgical Fear Scale | Baseline
  The Surgical Fear Scale, consisting of eight questions, is an 11-point Likert-type scale and is scored between 0 and 10. It consists of two sub-dimensions measuring short-term fears (items 1-4) and long-term fears (items 5-8) regarding the source of fear. The items in the scale are evaluated as "0: I am not afraid at all" and "10: I am very afraid". Increasing scores indicate increasing fear.
State Anxiety Inventory | Baseline
  The inventory consists of four-degree evaluations ranging from "Not at all" to "Completely" in the Likert type. There are 20 items in the inventory, and the individual is required to define how he/she feels at a certain moment and under certain conditions, and to respond by taking into account his/her feelings about the situation he/she is in. High scores indicate high anxiety levels, and low scores indicate low anxiety levels.
Visual Analog Scale | Baseline
  The scale is graded as 0-10 cm long, with 0=no pain, 10=the most severe pain. It is applied by the individual marking a point corresponding to the level of pain they feel. The distance between the determined point and the lowest part of the line is evaluated in centimeters. The value found indicates the patient's pain level.

SECONDARY OUTCOMES:
Surgical Fear Scale | through study completion, an average of 1 year
  The Surgical Fear Scale, consisting of eight questions, is an 11-point Likert-type scale and is scored between 0 and 10. It consists of two sub-dimensions measuring short-term fears (items 1-4) and long-term fears (items 5-8) regarding the source of fear. The items in the scale are evaluated as "0: I am not afraid at all" and "10: I am very afraid". Increasing scores indicate increasing fear.
State Anxiety Inventory | through study completion, an average of 1 year
  The inventory consists of four-degree evaluations ranging from "Not at all" to "Completely" in the Likert type. There are 20 items in the inventory, and the individual is required to define how he/she feels at a certain moment and under certain conditions, and to respond by taking into account his/her feelings about the situation he/she is in. High scores indicate high anxiety levels, and low scores indicate low anxiety levels.
Visual Analog Scale | through study completion, an average of 1 year
  The scale is graded as 0-10 cm long, with 0=no pain, 10=the most severe pain. It is applied by the individual marking a point corresponding to the level of pain they feel. The distance between the determined point and the lowest part of the line is evaluated in centimeters. The value found indicates the patient's pain level.

CONTACTS AND LOCATIONS:
Overall Officials: Sukran Ertekin Pinar, Assoc. Prof. Dr., Principal Investigator — Cumhuriyet University
Locations (1):
- Sukran Ertekin Pinar, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.